CLINICAL TRIAL: NCT06147063
Title: A Phase I, Open-label, Randomized, Active-Controlled Study in Adults to Characterize the Safety and Immunogenicity of AZD9838 and AZD6563 Vaccine (ARTEMIS-C)
Brief Title: A Randomized Trial Evaluating a mRNA-VLP Vaccine's Immunogenicity and Safety for COVID-19
Acronym: ARTEMIS-C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D8670C00001
Record Dates: First submitted 2023-11-24; First posted 2023-11-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; mRNA vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm 1: dosage 1 of AZD9838 18 to 64 years of age (Experimental): Participants will receive 1 intramuscular dose of AZD9838.
  Interventions: Biological: AZD9838
- Arm 2: dosage 2 of AZD9838 18 to 64 years of age (Experimental): Participants will receive 1 intramuscular dose of AZD9838.
  Interventions: Biological: AZD9838
- Arm 3: licensed mRNA vaccine 18 to 64 years of age (Active Comparator): Participants will receive 1 intramuscular dose of the licensed mRNA vaccine.
  Interventions: Biological: Licensed mRNA vaccine
- Arm 4: dosage 1 of AZD6563 18 to 64 years of age (Experimental): Participants will receive 1 intramuscular dose of AZD6563.
  Interventions: Biological: AZD6563
- Arm 5: dosage 2 of AZD6563 18 to 64 years of age (Experimental): Participants will receive 1 intramuscular dose of AZD6563.
  Interventions: Biological: AZD6563
- Arm 6: dosage 1 of AZD6563 65 years of age and older (Experimental): Participants will receive 1 intramuscular dose of AZD6563.
  Interventions: Biological: AZD6563
- Arm 7: dosage 2 of AZD6563 65 years of age and older (Experimental): Participants will receive 1 intramuscular dose of AZD6563.
  Interventions: Biological: AZD6563
- Arm 8: licensed mRNA vaccine 65 years of age and older (Active Comparator): Participants will receive 1 intramuscular dose of the licensed mRNA vaccine.
  Interventions: Biological: Licensed mRNA vaccine

INTERVENTIONS:
Biological: AZD9838 — Intramuscular (IM) injection.
  Arms: Arm 1: dosage 1 of AZD9838 18 to 64 years of age; Arm 2: dosage 2 of AZD9838 18 to 64 years of age
Biological: Licensed mRNA vaccine — Intramuscular (IM) injection.
  Arms: Arm 3: licensed mRNA vaccine 18 to 64 years of age; Arm 8: licensed mRNA vaccine 65 years of age and older
Biological: AZD6563 — Intramuscular (IM) injection.
  Arms: Arm 4: dosage 1 of AZD6563 18 to 64 years of age; Arm 5: dosage 2 of AZD6563 18 to 64 years of age; Arm 6: dosage 1 of AZD6563 65 years of age and older; Arm 7: dosage 2 of AZD6563 65 years of age and older

SUMMARY:
The purpose of this study is to characterize the safety and immunogenicity of AZD9838 and AZD6563 when administered as a single dose vaccination against SARS-CoV-2 in adults.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized, active-controlled study to assess the safety and immunogenicity of 2 dosages of AZD9838 and 2 dosages of AZD6563 compared with a licensed SARS-CoV-2 mRNA vaccine in approximately 240 healthy participants. AZD6563 will be assessed in adults 18 years of age and older. AZD9838 will be assessed in adults 18 to 64 years of age only.

The duration of each participant's involvement in the study will be approximately 12 months following administration of study vaccination.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥ 18 years at the time of signing informed consent.
* Self-reported History of SARS-CoV-2 infection at least 6 months prior to study vaccination AND/OR prior completion of primary series vaccination against COVID-19, with the final dose received at least 6 months prior to study vaccination
* Negative SARS-CoV-2 RT-PCR test at Visit 1
* Body mass index (BMI) of <35 kg/m2 at screening
* Medically stable - according to the judgement of the investigator, hospitalization within the study is not anticipated and participant is likely to remain in the study through the end of the protocol specified follow-up.

Key Exclusion Criteria:

* Acute illness/infection on day prior or day of dosing
* History of hypersensitivity to any component of the study vaccination, severe adverse reaction associated with a vaccine and/or severe allergic reaction
* Positive COVID-19 test result within 6 months of Visit 1
* Receipt of licensed, authorized, or investigational COVID-19 vaccines in the 6 months prior to administration of study intervention or expected receipt through completion of Visit 5.
* Receipt of any COVID-19 monoclonal antibody (licensed or investigational) within 3 months or receipt of immunoglobulin (non-COVID related) or blood products within 6 months prior to administration of study intervention, or expected receipt during the study
* Receipt of any licensed or investigational vaccine (other than licensed influenza vaccines or non-study COVID-19 vaccines) within 30 days prior to Visit 1 or expected receipt prior to completion of Visit 4. Licensed influenza vaccines are permitted beginning > 14 days before and > 14 days after administration of study intervention.
* Previous history of myocarditis or pericarditis
* Woman who are pregnant, lactating, or of child-bearing potential and not using a contraception or abstinence from at least 4 weeks prior to study vaccination and until at least 6 months after study vaccination
* Lab values above ULN (Serum creatinine, AST, ALT), below LLN (hemoglobin, WBC, Platelet count) or any lab value that in the opinion of the investigator is clinically significant or might confound analysis of the study results. Participants with laboratory values outside of the normal range may have the abnormal test repeated within the screening window and if the values are normal, then the participant can be randomized. If the repeated value remains outside of the normal range but it is not felt to be clinically significant by the Investigator, the case can be discussed with the AstraZeneca study physician and if they both agree the value is not clinically significant, the participant can be randomized
* History of malignancy within 5 years (treated non-melanoma skin cancer and locally treated cervical cancers allowed)
* Known or suspected congenital or acquired immunodeficiency
* Known or suspected autoimmune conditions as determined by history and /or physical examination
* Active infection with hepatitis B or C
* Troponin I levels above the normal range at the screening visit
* History of hypersensitivity to kanamycin or any aminoglycoside antibiotics (eg, neomycin, streptomycin, tobramycin, and gentamicin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of immediate unsolicited adverse events (AE) | Within 30 minutes post vaccination
  Number of participants who experienced immediate unsolicited AEs within 30 minutes post vaccination.
Incidence of solicited adverse reactions (AR) | Through 7 days post vaccination.
  Number of participants who experienced injection site and systemic solicited ARs through 7 days post vaccination.
Incidence of unsolicited adverse events (AE) | Through 28 days post vaccination.
  Number of participants who experienced unsolicited AEs through 28 days post vaccination.
Incidence of serious adverse events (SAE) | Through 12 months post vaccination
  Number of participants who experienced SAEs through 12 months post vaccination.
Incidence of medically attended adverse events (MAAE) | Through 12 months post vaccination
  Number of participants who experienced MAAEs through 12 months post vaccination.
Incidence of adverse events of special interest (AESI) | Through 12 months post vaccination
  Number of participants who experience AESIs through 12 months post vaccination.
Geometric mean titer (GMT) for SARS-CoV-2 ancestral strain neutralizing antibodies | Day 29
  GMT for SARS-CoV-2 ancestral strain neutralizing antibodies
Geometric mean titer (GMT) for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies | Day 29
  GMT for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies
Geometric mean titer (GMT) for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies | Day 29
  GMT for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies
Geometric mean fold rise (GMFR) for SARS-CoV-2 ancestral strain neutralizing antibodies | Day 1 to Day 29
  GMFR for SARS-CoV-2 ancestral strain neutralizing antibodies
Geometric mean fold rise (GMFR) for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies | Day 1 to Day 29
  GMFR for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies
Geometric mean fold rise (GMFR) for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies | Day 1 to Day 29
  GMFR for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies
Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 ancestral strain | Day 1 to Day 29
  Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 ancestral strain, defined as GMFR >=4 from baseline
Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron BA.4/5 | Day 1 to Day 29
  Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron BA.4/5, defined as GMFR >=4 from baseline
Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron XBB.1.5 | Day 1 to Day 29
  Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron XBB.1.5, defined as GMFR >=4 from baseline

SECONDARY OUTCOMES:
Geometric mean titer (GMT) for SARS-CoV-2 ancestral strain neutralizing antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 ancestral strain neutralizing antibodies by visit.
Geometric mean titer (GMT) for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies by visit.
Geometric mean titer (GMT) for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 ancestral strain neutralizing antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 ancestral strain neutralizing antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 Omicron BA.4/5 neutralizing antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 Omicron XBB.1.5 neutralizing antibodies by visit.
Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 ancestral strain | Day 1 to Day 360
  Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 ancestral strain, defined as GMFR >=4 from baseline by visit.
Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron BA.4/5 | Day 1 to Day 360
  Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron BA.4/5, defined as GMFR >=4 from baseline by visit.
Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron XBB.1.5 | Day 1 to Day 360
  Proportion of participants with neutralizing antibody seroresponse against SARS-CoV-2 Omicron XBB.1.5, defined as GMFR >=4 from baseline by visit.
Geometric mean titer (GMT) for SARS-CoV-2 ancestral strain S protein binding antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 ancestral strain S protein binding antibodies by visit.
Geometric mean titer (GMT) for SARS-CoV-2 Beta variant S protein binding antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 Beta variant S protein binding antibodies by visit.
Geometric mean titer (GMT) for SARS-CoV-2 Delta variant S protein binding antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 Delta variant S protein binding antibodies by visit.
Geometric mean titer (GMT) for SARS-CoV-2 Omicron subvariant S protein binding antibodies | Day 1 to Day 360
  GMT for SARS-CoV-2 Omicron subvariant S protein binding antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 ancestral strain S protein binding antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 ancestral strain S protein binding antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 Beta variant S protein binding antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 Beta variant S protein binding antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 Delta variant S protein binding antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 Delta variant S protein binding antibodies by visit.
Geometric mean fold rise (GMFR) for SARS-CoV-2 Omicron subvariant S protein binding antibodies | Day 1 to Day 360
  GMFR for SARS-CoV-2 Omicron subvariant S protein binding antibodies by visit.
Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 ancestral strain | Day 1 to Day 360
  Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 ancestral strain by visit.
Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 Beta variant | Day 1 to Day 360
  Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 Beta variant by visit.
Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 Delta variant | Day 1 to Day 360
  Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 Delta variant by visit.
Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 Omicron subvariant | Day 1 to Day 360
  Proportion of participants with S protein binding antibody seroresponse against SARS-CoV-2 Omicron subvariant by visit.
Geometric mean response of S-specific Th1 and Th2 by cytokine-producing T cells by phenotype | Day 1 to Day 180
  Geometric mean response of S-specific Th1 and Th2 by cytokine-producing T cells by phenotype as measured by an intracellular cytokine staining assay over time.
Incidence and titer of H. pylori and human anti-ferritin antibodies | Day 1 to Day 360
  Incidence and titer of H. pylori and human anti-ferritin antibodies over time.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Long Beach, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Chicago, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home